CLINICAL TRIAL: NCT05365854
Title: Comparison of Hemodynamic Effects of Two Modalities of Alveolar Recruitment Maneuvers in Intensive Care Unit Patients Under Mechanical Ventilation. A Pilot Physiological Study
Brief Title: Hemodynamic Effects of Two Modalities of Alveolar Recruitment Maneuvers - ICU Patients
Acronym: CHARM-ICU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: RBPH 2021 GODET 3 (Charm ICU)
Record Dates: First submitted 2022-04-19; First posted 2022-05-09 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-02

CONDITIONS: Cardiac Output; Hemodynamic Optimization; Monitoring Blood Pressure; Stroke Volume; Mechanical Ventilation; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous positive airway pressure (CPAP) then extended sigh (Active Comparator): Patients assigned to this group will receive a CPAP ARM (40cmH2O during 50 seconds), followed by a 10-minute pause corresponding to a period of return to basal state.
  Then an ARM by extended sigh (e-sigh) also 50 seconds (driving pressure at 10cmH2O and successive PEEP levels at 10, 15, 20, 25 and 30cmH2O, with respiratory frequency fixed at 30/min in controlled pressure).
  Hemodynamic (blood pressure, cardiac output, stroke volume) and ventilatory measurements will be performed the last 10 seconds of each recruitment maneuver.
  Interventions: Procedure: Alveolar Recruitment Maneuver (ARM)
- extended sigh then continuous positive airway pressure (CPAP) (Active Comparator): Patients assigned to this group will receive an ARM by extended sigh (e-sigh) during 50 seconds (driving pressure at 10cmH2O and successive PEEP levels at 10, 15, 20, 25 and 30cmH2O, with respiratory frequency fixed at 30/min in controlled pressure), followed by a 10-minute pause corresponding to a period of return to basal state.
  Then they receive a CPAP ARM (40cmH2O during 50 seconds). Hemodynamic (blood pressure, cardiac output, stroke volume) and ventilatory measurements will be performed the last 10 seconds of each recruitment maneuver.
  Interventions: Procedure: Alveolar Recruitment Maneuver (ARM)

INTERVENTIONS:
Procedure: Alveolar Recruitment Maneuver (ARM) — When patient is under general anesthesia, an arterial catheter is placed for cardiac output and stroke volume (SV) monitoring. To avoid pre-load dependency bias, the blood volume will be optimized. A 250mL fluid-challenge of a balanced crystalloid solution is administered under cover of the SV monitoring. If SV variation is greater than 10%, a new fluid-challenge is performed to obtain a reference SV, corresponding to the patient's optimal blood volume.The patient is then "pre-load independent".
  Then, patients will be randomized into two groups: a first group will receive a CPAP ARM: 40 cmH2O for 50 seconds, followed by a 10-minute break corresponding to a period of return to basal state; then an extended sigh ARM (e-sigh) also lasting 50seconds (driving pressure: 10cmH2O and successive PEEP levels at 10,15,20,25 and 30cmH2O, a respiratory rate set at 30/min in controlled pressure - 5cycles at each PEEP level); a second group will receive the same two ARM modalities in reverse order.

SUMMARY:
The objective of this study was to investigate the hemodynamic effects of two alveolar recruitment maneuver strategies in critical care patients with acute respiratory distress syndrome.

DETAILED DESCRIPTION:
Critical care patients are at risk of significant variations in blood volume due to long intervention times, major bleeding or serious pathological conditions, requiring invasive hemodynamic monitoring in routine practice, in order to optimize blood volume and ensure adequate perfusion of the organs, throughout their care.

The installation of an arterial catheter allows continuous monitoring of blood pressure and the realization of blood tests if necessary.

The installation of a central venous line allows the administration of anesthetic drugs and vasopressors as well as an accurate hemodynamic evaluation by transpulmonary thermodilution, which is the most commonly used monitoring in these situations.

After hemodynamic optimization following the monitoring data, the patient will be randomized to one of the two Alveolar Recruitment Maneuver (ARM) order strategies. Mechanical ventilation will be standardized according to current international recommendations (tidal volume between 6 mL.kg-1 and 8 mL.kg-1 of theoretical ideal weight (TIP) for patients with Acute Respiratory Distress Syndrome (ARDS); PEEP equal to 6 cmH2O). Hemodynamic and ventilatory data will be collected (baseline).

The successive realization of the two ARM will then be carried out with collection of the hemodynamic and ventilatory data during the last 10 seconds of each ARM. Between each ARM, conventional ventilation will be resumed for 10 minutes in order to observe a wash-out period, and to allow a return to the baseline state. Data will also be collected as before.

After these measurements have been taken, all management will be left to the discretion of the practitioner caring for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Patient under general anesthesia
* Intubated patient under controlled invasive mechanical ventilation
* Patient with invasive hemodynamic monitoring allowing monitoring of cardiac output and stroke volume
* Patient sufficiently sedated (BIS between 40 and 60) and/or curarized (TOF < 2/4 at the orbicularis) to avoid inspiratory effort
* Patient optimized on the hemodynamic level, in particular with regard to blood volume, following the data from hemodynamic monitoring and the recommendations of the French Society of Anesthesia and Resuscitation (RFE SFAR 2013 - Perioperative Vascular Filling Strategy)
* Patient covered by a Social Security plan
* Consent of close relatives or trusted person (if present)
* Patient admitted in polyvalent resuscitation within the Peri-Operative Medicine Unit of Clermont-Ferrand hospital suffering from respiratory distress syndrome for less than 24 hours

Exclusion Criteria:

* Contraindication to the use of cardiac output measurement by transpulmonary thermodilution
* Cardiac arrhythmia
* Severe valvulopathy
* Contraindication to the use of the Analysis of pulmonary aeration will be performed using the non-invasive technique of electrical impedance tomography with the placement of an electrode belt on the patient's chest. Values will be recorded with this belt :

technique

* Left ventricular ejection fraction (LVEF) < 45% and/or right ventricular failure
* History of pulmonary lobectomy and/or pneumectomy and/or known emphysema
* Patient with restrictive or obstructive lung disease
* Body mass index (BMI) < 16.5 or > 30 kg.m-2
* Pregnancy
* Major under legal protection (guardianship, curators, safeguard of justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is the change in cardiac output during the last 10 seconds of each ARM modality from its baseline value (determined after hemodynamic optimization and before the procedure was performed) | During procedure (last 10 seconds of each ARM modality)
  Cardiac output (l/min) will be measured by invasive monitoring during the last 10 seconds of each recruitment maneuver

SECONDARY OUTCOMES:
The secondary outcome measures are the evaluation of standard hemodynamic monitoring data | During procedure (last 10 seconds of each ARM modality)
  During the last 10 seconds of the recruitment maneuver, standard hemodynamic monitoring data will be recorded :
  blood pressure (mmHg) mean arterial pressure (mmHg)
Standard hemodynamic monitoring data | During procedure (last 10 seconds of each ARM modality)
  heart rate
Invasive hemodynamic monitoring data | During procedure (last 10 seconds of each ARM modality)
  stroke volume (ml/min)
Invasive hemodynamic monitoring data | During procedure (last 10 seconds of each ARM modality)
  change in stroke volume
Standard ventilatory monitoring data | During procedure (last 10 seconds of each ARM modality)
  tidal volume (ml)
Standard ventilatory monitoring data | During procedure (last 10 seconds of each ARM modality)
  positive end-expiratory pressure (PEEP), peak pressure, plateau inspiration pressure, driving pressure,
Standard ventilatory monitoring data | During procedure (last 10 seconds of each ARM modality)
  respiratory rate
Standard ventilatory monitoring data | During procedure (last 10 seconds of each ARM modality)
  inspired oxygen fraction
Standard ventilatory monitoring data | During procedure (last 10 seconds of each ARM modality)
  compliance of the respiratory system
Electrical impedance tomography data | During procedure (last 10 seconds of each ARM modality)
  Analysis of pulmonary aeration will be performed using the non-invasive technique of electrical impedance tomography with the placement of an electrode belt on the patient's chest. Values will be recorded with this belt :
  Tidal Impedance Variation (TIV)
Electrical impedance tomography data | During procedure (last 10 seconds of each ARM modality)
  Analysis of pulmonary aeration will be performed using the non-invasive technique of electrical impedance tomography with the placement of an electrode belt on the patient's chest. Values will be recorded with this belt :
  Center Of Ventilation (COV) and Global Inhomogeneity index (GI)
Electrical impedance tomography data | During procedure (last 10 seconds of each ARM modality)
  Analysis of pulmonary aeration will be performed using the non-invasive technique of electrical impedance tomography with the placement of an electrode belt on the patient's chest. Values will be recorded with this belt :
  Regional Ventilation Delay (RVD)
Electrical impedance tomography data | During procedure (last 10 seconds of each ARM modality)
  Analysis of pulmonary aeration will be performed using the non-invasive technique of electrical impedance tomography with the placement of an electrode belt on the patient's chest. Values will be recorded with this belt :
  End Expiratory Lung Impedance (EELI)
Electrical impedance tomography data | During procedure (last 10 seconds of each ARM modality)
  Analysis of pulmonary aeration will be performed using the non-invasive technique of electrical impedance tomography with the placement of an electrode belt on the patient's chest. Values will be recorded with this belt :
  percentages of overdistended and atelectasis areas
The secondary outcome measures are the evaluation of paraclinical data | During procedure (last 10 seconds of each ARM modality)
  During the last 10 seconds of the recruitment maneuver, capnography will be recorded
The secondary outcome measures are the evaluation of paraclinical data | During procedure (last 10 seconds of each ARM modality)
  During the last 10 seconds of the recruitment maneuver, pulse oxygen saturation (SpO2) will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- CHU, Clermont-Ferrand, France